CLINICAL TRIAL: NCT06498518
Title: PRIMUS 006 - A Phase II Trial of Gemcitabine, Pembrolizumab and IMM-101 as First Line Treatment in Patients With Metastatic Pancreatic Cancer
Brief Title: A Trial of Gemcitabine, Pembrolizumab and IMM-101 as First Line Treatment in Patients With Metastatic Pancreatic Cancer
Acronym: PRIMUS006
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: One of the pharmaceutical partners (Immodulon) went into administration, the company which bought the assets confirmed to the study team on 23rd May 2025 they were not in position to support the study. Study terminated early
Sponsor: Karen Carty (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); University of Glasgow (Other)
Responsible Party: Sponsor-Investigator, Karen Carty, Mrs, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIMUS006-2022
Record Dates: First submitted 2024-07-02; First posted 2024-07-12 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — IMM-101; pembrolizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMM-101, Pembrolizumab and Gemcitabine (Experimental): IMM-101: will be administered at a dose of 1mg intra-dermal (ID) between 2 to 7 days prior to first cycle of pembrolizumab (MK-3475)/ gemcitabine then 1mg ID on day 8 of cycle 1, 1mg on day 1 of cycle 2, 1mg on day 8 of cycle 3 then 1mg on day 8 of each cycle thereafter.
  Pembrolizumab (MK-3475): will be administered at a dose of 200mg by IV infusion every 3 weeks starting from cycle 1, day 1.
  Gemcitabine: will be administered at a dose of 1000mg/m2 by IV infusion on day 1 and day 8 of every 3 week-cycle starting from cycle 1, day 1.
  Each cycle is 3 weeks
  Interventions: Drug: IMM-101, Pembrolizumab, Gemcitabine

INTERVENTIONS:
Drug: IMM-101, Pembrolizumab, Gemcitabine — Patients will receive IMM-101, Pembrolizumab, Gemcitabine on a 3 week cycle

SUMMARY:
Trial to investigate if the addition of two novel immunotherapy agents in combination with a chemotherapy agent can reduce the size of the cancer and how long they can delay the growth of the cancer in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The PRIMUS-006 study is a study for first line metastatic pancreatic cancer patients with Eastern Co-operative Oncology Group (ECOG) performance status 1, who are not sufficiently fit to tolerate a combination treatment regimen of two or more cytotoxic chemotherapy agents in the opinion of the investigator. The study is a single arm phase II signal seeking trial of gemcitabine + pembrolizumab + IMM-101 (a heat inactivated mycobacterium, immune modulator) using objective response rate as the primary endpoint

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged > or = 18 years for age
2. Patient has given written informed consent to participate in the trial
3. Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma or its variants
4. Patient has been enrolled in the Precision-Panc Master Protocol and their tissue has been deemed suitable for Next Generation Sequencing (NGS) analysis.
5. No prior systemic anti-cancer therapy for metastatic pancreatic cancer. Patients may have received prior pre-, peri-, or post-operative systemic anti-cancer therapy for operable disease with curative intent provided that the last dose of systemic anti-cancer therapy was completed > 6 months before the recurrent disease was documented
6. ECOG performance status 1, but not sufficiently fit to potentially tolerate treatment with a combination treatment regimen consisting of two or more cytotoxic chemotherapy agents in the opinion of the investigator.
7. Measurable disease by RECIST 1.1.
8. Estimated life expectancy > 3 months.
9. Adequate haematological and biochemical function.
10. Willingness to comply with study procedures including administration of study therapies.
11. Females of childbearing potential must have a negative pregnancy test within 72 hours of the first dose of study treatment and agree to use highly effective contraceptive measures during the study and for 6 months after the last administration of the study drug.
12. Male patients with partners of childbearing potential must agree to use highly effective contraceptive measures during the study and for 6 months after the last administration of the study drug
13. Patients with a history of Hepatitis C Virus (HCV) infection are eligible for the study if HCV viral load is undetectable at screening. Patients who have been treated for HCV infection must have completed curative anti-viral therapy at least 4 weeks before registration to the trial.
14. Patients who are hepatitis B positive will be eligible as long as they meet the following criteria:

14.1. Patients who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks and have an undetectable HBV viral load before registration to the trial 14.2. Patients should remain on anti-viral therapy throughout study treatment and follow local guidelines for HBV anti-viral therapy post-completion of study treatment

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Patients with cardiovascular disease defined as Stage II to IV congestive heart failure (CHF) as determined by the New York Heart Association (NYHA) classification system, or history of myocardial infarction (MI), or cardiac arrhythmia associated with haemodynamic instability, or unstable angina, or cerebral vascular accident, or transient ischemia, if any have occurred within the previous 12 months prior to study treatment.
3. Any other serious medical or psychiatric disorder that would be, in the opinion of the investigator, a contra-indication to either the trial procedures or to therapy with gemcitabine, IMM-101 or pembrolizumab.
4. Any prior therapy with IMM-101 or an immune checkpoint inhibitor.
5. Major surgery within 28 days of starting study treatment and patients must have recovered from any effects of major surgery.
6. Patients with a known hypersensitivity to gemcitabine, IMM-101, or pembrolizumab or any of the excipients of the products, including patients who have previously experienced an allergic reaction to any mycobacterial product.
7. Current or prior use of immunosuppressive medication within 14 days before the first dose of IMM-101 or pembrolizumab. The following are exceptions to this criterion:

   7.1. Intranasal, inhaled, or topical steroids; or local steroid injections (e.g., intra-articular injection) 7.2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisolone or equivalent 7.3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) and chemotherapy-induced nausea and vomiting
8. History of allogenic organ transplant.
9. Previous severe or life-threatening skin adverse reaction with other immune-stimulatory anticancer agents.
10. Active autoimmune disorders, or prior documented severe autoimmune or inflammatory disorders requiring immunosuppressive treatment in the last 2 years (including inflammatory bowel disease [e.g., colitis, Crohn's disease], diverticulitis with the exception of diverticulosis, coeliac disease, irritable bowel syndrome, or other serious gastrointestinal chronic conditions associated with diarrhoea); systemic lupus erythematosus; Wegener syndrome (granulomatosis with polyangiitis), Graves' disease; rheumatoid arthritis, hypophysitis, uveitis or other evidenced autoimmune disorders. The following are exceptions to this criterion:

    10.1. Patients with vitiligo or alopecia 10.2. Diabetes mellitus type I or resolved childhood asthma/atopy 10.3. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement 10.4. Any chronic skin condition that does not require systemic therapy 10.5. Patients with coeliac disease controlled by diet alone
11. History of (non-infectious) interstitial lung disease or pneumonitis that required steroids or current pneumonitis.
12. Patients with an active infection requiring systemic therapy.
13. Concurrent active Hepatitis B (defined as HBsAG positive and/or detectable HBV/DNA) or Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
14. History of (non-infectious) interstitial lung disease or pneumonitis that required steroids or current pneumonitis.
15. Patients with an active infection requiring systemic therapy.
16. Receipt of the last dose of an approved (marketed) anticancer therapy (chemotherapy, targeted therapy, biologic therapy, monoclonal antibodies, etc.) or radiotherapy within 28 days or 5 half-lives, whichever is the longest, prior to the first dose of study treatment.
17. Received prior radiotherapy within 2 weeks of the start of the study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-Central Nervous System (CNS) disease.
18. Other malignancy within 3 years except for non-invasive malignancies such as cervical carcinoma in situ, non-melanoma carcinoma of the skin, or ductal carcinoma in situ of the breast that has/have been surgically cured or treated/biochemically-stable, organ-confined prostate cancer (patients can remain on treatment for this indication as long as not contraindicated with study treatment).
19. Receipt of a live attenuated vaccine within 30 days prior to the first dose of study th

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Measured every 6 weeks by CT scan(most patients will receive 3-4 CT scans over 24 weeks)
  The proportion of patients achieving an objective response, defined by RECIST 1.1, measured using CT scans for radiological assessment of disease until disease progression

SECONDARY OUTCOMES:
Progression Free Survival | At time of progression (estimated to be between 3 and 6 months)
  Progression Free survival as measured from date of registration to progression or death (from any cause)
Safety and Tolerability of Gemcitabine in combination with IMM-101 and Pembrolizumab | Measured during combination treatment and for up to at least 30 days after the last dose of study therapies. In addition, immune mediated adverse events that occur up to 90 days after the last dose of pembrolizumab
  Occurrence and Frequency of grade 1-5 adverse events measured using NCI CTCAE Version 5
Overall Survival | From date of registration until date of death from any cause ( estimated to be between 6-12 months)
  Survival will be measured from the date of registration and include all causes of death

CONTACTS AND LOCATIONS:
Overall Officials: David Chang, Study Chair — University of Glasgow; Jeff Evans, Study Chair — University of Glasgow
Locations (6):
- United Kingdom (6):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - University Hospitals Coventry & Warwickshire, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free London Hospital, London
  - Royal Marsden Hospital, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, once the study report has been written and published the anonymised clinical data will be available via requests to the Trial Management Group and Co-ordinating Clinical Trials Unit
Supporting Information: Study Protocol, CSR
Time Frame: After publication of the study
Access Criteria: Available via request to the Trial Management Group and Co-ordinating Clinical Trials Unit